CLINICAL TRIAL: NCT04786925
Title: Strategies for Improving the Quality of Life of Pre-senior and Senior Populations Based on Precision Nutrition (Proyecto Nutriprecisión)
Brief Title: Precision Nutrition Strategies for Improving the Quality of Life of Pre-senior and Senior Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Principal Investigator, Itziar Abete, Principal Investigator, Clinica Universidad de Navarra, Universidad de Navarra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NUTRIPRECISION
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Overweight or Obesity
Keywords: Obesity; Health status; Insulin resistance; Hypertension; Lipid profile; Gastrointestinal health; Cognitive capacity; Life quality; Healthy ageing; Lifestyle intervention; Precision nutrition; Mediterranean diet; Eating behaviour; Physical activity; Oxidative stress; Inflammation; Functional ability; Nutrition education
MeSH Terms: conditions — Overweight; Obesity; Insulin Resistance; Hypertension; Feeding Behavior; Motor Activity; Inflammation

STUDY DESIGN:
Intervention Model Description: The participants are randomly assigned to Control or NUTRIPRECISION strategy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control diet (Placebo Comparator): A conventional diet based on the current Spanish Mediterranean dietary guidelines: Spanish Society of Community Nutrition (SENC).
  Interventions: Other: Control diet
- Nutriprecision diet (Experimental): A Mediterranean, balanced diet based on the inclusion of precision foods designed and developed within the framework of Nutriprecision project. A mobile application to empower and support the management of the dietary prescription. A digital tool for cognitive stimulation.
  Interventions: Other: Nutriprecision diet

INTERVENTIONS:
Other: Control diet — Control diet: A Mediterranean conventional diet based on the current dietary guidelines of the Spanish Society of Community Nutrition (SENC). Participants were strongly advised to use the Healthy Eating Plate (Harvard) to structure and prepare the main meals (lunch and dinner). In this way, at least ½ of the plate should be composed of vegetables, ¼ of lean protein, and ¼ of low glycemic index carbohydrates. The diet encourages participants to eat 5 times/day (breakfast, lunch, dinner, and two snacks). Overall, the control diet was based on high consumption of vegetables and fruits, whole grains, healthy fats (olive oil), and healthy proteins (legumes, fish, and lean meat). There was not energy restriction in the control diet.
  Arms: Control diet
Other: Nutriprecision diet — Nutriprecision diet: a Mediterranean balanced diet based on the inclusion of precision foods designed according to the particularities of the senior population. The selected precision foods were a) fruit compote, b) smoothie, c) extruded meat product, d) wholemeal bread, e) wholemeal biscuit and f) microwaveable deep-frozen vegetable products. The diet encourages participants to eat 5 times/day with a conventionally balanced distribution of macronutrients (50% of the total caloric value from carbohydrates, 20% from proteins, and 30% from lipids). There was not energy restriction, although the energy requirements of the participants were adjusted to a BMI of 25 kg/m2 to avoid an overestimate of calorie intake. A mobile application designed and developed to provide volunteers with information about follow-up visits, the assigned diet, recommendations, and messages to motivate them during the intervention. A digital tool for cognitive stimulation.
  Arms: Nutriprecision diet

SUMMARY:
The number and proportion of people aged 60 years old and over is increasing worldwide. Ageing is characterized by a progressive loss of physiological integrity, leading to impaired function and increased vulnerability to death. This deterioration is the primary risk factor for major chronic diseases including diabetes, cardiovascular disease, and neurodegenerative disorders.

The incidence of chronic conditions frequently rises sharply with age, after long exposure to unhealthful lifestyles involving the consumption of unhealthy diets and physical inactivity. Consequently, integrated dietary strategies and actions are required to promote healthy ageing and target major causes of morbidity and mortality in senior populations.

The promising field of precision nutrition is rising as a therapeutic approach that aims to design tailored dietary interventions to prevent and manage chronic diseases. Indeed, precision nutrition approaches contemplate the interindividual heterogeneity caused by genetic/epigenetic dissimilarities, individual facets such as age and gender, the lifestyle and environmental exposome diversity, microbiome variations, and singular behavioral/psychological features.

On the other hand, the inclusion of potentially bioactive compounds and functional foods as promoters of healthy aging within personalised dietary patterns could be an effective strategy to delay the aging process and age-related chronic diseases.

One of the main limitations of a dietary prescription is the lack of compliance, due to the complexity of the prescription itself and/or the lack of commitment of the individual. The inclusion of digital tools to empower and motivate individuals and to support them in the management of the dietary strategy could overcome this limitation.

With this background, the general objective of this investigation is to design precision nutritional strategies based on the inclusion of functional foods and digital tools for preventing age-related chronic diseases in pre-senior and senior populations. Additionally, this study proposes alternative tools for cognitive assessments increasing the accessibility to cognitive assessment tools for this population as well as an innovative digital tool for cognitive stimulation which is personalized, monitored, and evidence-based.

DETAILED DESCRIPTION:
This study is designed as a 12-week, randomized parallel intervention trial, with two arms: 1) Control group, who follows a control diet based on the current dietary guidelines of the Spanish Society of Community Nutrition (SENC) using the Healthy Eating Plate method (Harvard), and 2) Nutriprecision Group, which were instructed to follow the Nutriprecision diet based on the inclusion of digital tools and functional foods, whose postprandial effects were previously evaluated by randomized, cross-over, double-blind studies in senior subjects in the Centre for Nutrition Research (UNAV) and IMDEA-ALIMENTACIÓN. The incremental area under the curve (iAUC) for glucose and insulin was calculated for all designed foods and was compared with their reference products. Additionally, lipid profile and satiety were measured at fasting and at 15, 30, 45, 60, 90, and 120 min after starting the food intake. In all these studies, the reference and test foods were administered once in random order, with a wash-out period between 7 days and 14 days among assays.

This multi-centric study was carried out in the Nutrition Intervention Unit of the Centre for Nutrition Research in the University of Navarra and the Nutritional and Clinical Trials Unit in IMDEA-ALIMENTACIÓN by qualified professionals (nurse, doctor-dietician, dieticians, pharmacists).

A total of five visits had been established along with the 12-weeks trial: 1) study information and screening; 2) day 0: start of the intervention; 3) day 28: group session (control group)/follow-up visit (Nutriprecision group); 4) day 56: group session (control group)/follow-up visit (Nutriprecision group) and 5) day 84: end of the intervention.

At the start and finish days of the study, participants visited the Nutrition Intervention Unit or the Clinical Trials Unit in a fasting state. Participants were instructed to collect the first-morning urine sample. Additionally, volunteers from the University of Navarra self-collected fecal samples at baseline using OMNIgene.GUT kits from DNA Genotek. Volunteers were also informed of a digital-based procedure for cognitive assessment and other digital tools available depending on the assigned intervention (experimental VS control).

Blood samples were drawn by venipuncture after a 12 h overnight fast in a clinical setting. After 10 minutes of rest and having answered the Mini Nutritional Assessment (MNA) and the Mini-Mental State Examination (MMSE) questionnaires, blood pressure was measured. Later, anthropometric measurements and body composition analysis were performed. Global cognitive performance was also assessed by the Guttmann NeuroPersonalTrainer platform. The duration of these visits was approximately 1 hour.

On the 28th and 56th study days, participants assigned to the control group attended online group sessions and received intensive education and advice to increase the adherence to the dietary strategy. Sessions consisted of informative talks about the prescribed dietary pattern, food label use, seasonal shopping lists, meal plans and recipes, physical activity and exercise recommendations, sleep habits, etc. Contrary, participants allocated to the Nutriprecision group attended in person visits with the dieticians, to evaluate the adherence to the assigned nutritional treatment. Additionally, anthropometric, body composition, and blood pressure measurements were assessed. Participants were also asked to fill different questionnaires about health status (SF-36 Health Survey), gastrointestinal symptoms (gastrointestinal symptoms rating scale, GSRT), dietary assessment (7-day recall), Mediterranean diet adherence (14-Item Mediterranean Diet Assessment Tool), physical activity (International Physical Activity Questionnaire, IPAQ) and drug therapy modifications. Moreover, the Nutriprecision group were asked to collect a sensory perception questionnaire and a food consumption record of the precision foods administered.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 50-80 years
* BMI >27 kg/m2
* One or more of the following risk factors:

  * Glucose ≥100 to ≤125 mg/dL or type 2 diabetes (independently of antidiabetic medication)
  * Hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg or under antihypertensive medication)
  * LDL-cholesterol ≥160 mg/dL independently of lipid-lowering therapy
  * HDL-cholesterol ≤40 mg/dL (men)/≤50 mg/dL (women), independently of lipid-lowering therapy
  * Triglycerides ≥160 mg/dL independently of lipid-lowering therapy
  * Waist Circumference ˃95 cm (men)/>82 cm (women), independently of lipid-lowering therapy
  * Sedentary behavior (AHA)*

Exclusion Criteria:

* Relevant functional or structural digestive abnormalities (malformations, angiodysplasia, active peptic ulcers, chronic inflammatory diseases, or malabsorption)
* Endocrine disorders (hyperthyroidism or uncontrolled hypothyroidism)
* Undergone surgical interventions with permanent sequelae (gastroduodenostomy)
* Pharmacological treatments with immunosuppressants, cytotoxic agents, systemic corticosteroids, or other drugs that could potentially cause hepatic steatosis or alteration of liver tests
* Active cancer in the last five years or under therapy
* Weight loss ≥3 kg in the last three months
* Instable drug therapy in the last three months
* Severe psychiatric disorders
* No autonomy
* Inability to follow the diet (food allergies, intolerances)
* Difficulties to follow scheduled visits

  * AHA Recommendations for Physical Activity in Adults: at least 150 minutes per week of moderate-intensity aerobic activity or 75 minutes per week of vigorous aerobic activity, or a combination of both, preferably spread throughout the week.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Change From Baseline General Health Status at 3 Months | 0 months and 3 months
  General health score encompassed twelve parameters, on a scale of 0 to 21, with higher scores indicating a worse overall health:
  * BMI
  * Waist Circumference
  * Glycosylated hemoglobin (HbA1C)
  * Total cholesterol
  * HDL-cholesterol
  * LDL-cholesterol
  * Triglycerides
  * Uric acid
  * Systolic Blood Pressure | Diastolic Blood Pressure
  * Gastrointestinal Health (GSRT)
  * Cognitive Function
  * Extra negative point if reducing medication

SECONDARY OUTCOMES:
Change From Baseline Weight at 3 Months | 0 months and 3 months
  Weight was measured by a digital scale
Baseline height | 0 months
  Height was recorded using a wall-mounted stadiometer (Seca 220, Vogel & Halke, Germany).
Change From Baseline Body Mass Index at 3 Months | 0 months and 3 months
  Body mass index was calculated using the standard formula: weight (kg)/height (m)2
Change From Baseline Fat Mass at 3 Months | 0 months and 3 months
  Fat mass was measured by Bioelectrical impedance analysis (BIA, SC-330, Tanita)
Change From Baseline Lean Mass at 3 Months | 0 months and 3 months
  Lean mass was measured by Bioelectrical impedance analysis (BIA, SC-330, Tanita)
Change From Baseline Waist Circumference at 3 Months | 0 months and 3 months
  Waist Circumference was measured by with a tape measure
Change From Baseline Hip Circumference at 3 Months | 0 months and 3 months
  Hip Circumference was measured by with a tape measure
Change From Baseline Systolic Blood Pressure at 3 Months | 0 months and 3 months
  Systolic Blood Pressure was measured using an automatic monitor device (Intelli Sense. M6, OMRON Healthcare, Hoofdorp, the Netherlands)
Change From Baseline Diastolic Blood Pressure at 3 Months | 0 months and 3 months
  Diastolic Blood Pressure was measured using an automatic monitor device (Intelli Sense. M6, OMRON Healthcare, Hoofdorp, the Netherlands)
Change From Baseline Serum Triglycerides at 3 Months | 0 months and 3 months
  Triglycerides were measured in fasting conditions
Change From Baseline Serum Total Cholesterol at 3 Months | 0 months and 3 months
  Total cholesterol was measured in fasting conditions
Change From Baseline Serum LDL-Cholesterol at 3 Months | 0 months and 3 months
  LDL-cholesterol was measured in fasting conditions
Change From Baseline Serum HDL-Cholesterol at 3 Months | 0 months and 3 months
  HDL-cholesterol was measured in fasting conditions
Change From Baseline Serum Uric Acid at 3 Months | 0 months and 3 months
  Uric acid was measured in fasting conditions
Change From Baseline Serum Glucose at 3 Months | 0 months and 3 months
  Glucose was measured in fasting conditions
Change From Baseline Serum Insulin at 3 Months | 0 months and 3 months
  Insulin was measured in fasting conditions
Change From Baseline Serum Glycosylated hemoglobin (HbA1C) at 3 Months | 0 months and 3 months
  Glycosylated hemoglobin (HbA1C) was measured in fasting conditions
Change From Baseline Serum Aspartate Aminotransferase at 3 Months | 0 months and 3 months
  Aspartate aminotransferase was measured in fasting conditions
Change From Baseline Serum Alanine Aminotransferase at 3 Months | 0 months and 3 months
  Alanine aminotransferase was measured in fasting conditions
Change From Baseline Serum Gamma-glutamyltransferase at 3 Months | 0 months and 3 months
  Gamma glutamyltransferase was measured in fasting conditions
Change From Baseline Physical Activity Level at 3 Months | 0 months and 3 months
  Physical activity was measured by the International Physical Activity Questionnaire (IPAQ)
Change From Baseline Dietary Intake at 3 Months | 0 months and 3 months
  Dietary intake was measured by a 7-day recall
Change From Baseline Mediterranean Diet Adherence at 3 Months | 0 months and 3 months
  Mediterranean diet adherence was measured by the 14-Item Mediterranean Diet Assessment Tool
Change From Baseline Health Status at 3 Months | 0 months and 3 months
  Health status was measured by the SF-36 Health Survey
Change From Baseline Gastrointestinal Symptoms at 3 Months | 0 months and 3 months
  Gastrointestinal symptoms were measured by the gastrointestinal symptoms rating scale, GSRT
Change From Baseline Sensory Perception of Precision Foods at 3 Months | 1 month and 3 months
  Sensory perception of precision foods was measured by the sensory perception questionnaire
Food Consumption of the Precision Foods | 1 month, 2 months and 3 months
  Food consumption of the precision foods was measured by a food consumption record
Change From Baseline Risk of Malnutrition at 3 Months | 0 months and 3 months
  Risk of malnutrition was measured by the Mini Nutritional Assessment (MNA) questionnaire
Change From Baseline Cognitive Impairment at 3 Months | 0 months and 3 months
  Cognitive impairment was measured by the Mini-Mental State Examination (MMSE) questionnaire
Change From Baseline Cognitive Function at 3 Months | 0 months and 3 months
  Cognitive function was measured by the Guttmann NeuroPersonalTrainer platform
Baseline Gut Microbiota Composition | 0 months
  Gut Microbiota Composition will be measured using OMNIgene.GUT kits from DNA Genotek
Usability of the digital tools | 3 months
  Usability will be measured using the System Usability Scale (SUS)
Baseline subjective hunger | Baseline
  Visual analogue scale rating in a scale from 0 to 100 mm, for the quantification of the perceived hunger before the experimental food intake
Postprandial subjective hunger | Up to 120 minutes
  Visual analogue scale rating in a scale from 0 to 100 mm, for the quantification of the perceived hunger measured at 15, 30, 45, 60, 90 and 120 minutes after the experimental food intake
Baseline subjective fullness | Baseline
  Visual analogue scale rating in a scale from 0 to 100 mm for the quantification of the perceived fullness before the experimental food intake
Postprandial subjective fullness | Up to 120 minutes
  Visual analogue scale rating in a scale from 0 to 100 mm, for the quantification of the perceived fullness measured at 15, 30, 45, 60, 90 and 120 minutes after the experimental food intake
Baseline subjective satiety | Baseline
  Visual analogue scale rating in a scale from 0 to100 mm for the quantification of the perceived satiety before the experimental food intake.
Postprandial subjective satiety | Up to 120 minutes
  Visual analogue scale rating in a scale from 0 to100 mm for the quantification of the perceived satiety measured at 15, 30, 45, 60, 90 and 120 minutes after experimental food intake
Baseline subjective desire to eat | Baseline
  Visual analogue scale rating in a scale from 0 to 100 mm for the quantification of the perceived desire to eat before the experimental food intake at baseline.
Postprandial subjective desire to eat | Up to 120 minutes
  Visual analogue scale rating in a scale from 0 to 100 mm for the quantification of the perceived desire to eat measured at 15, 30, 45, 60, 90 and 120 minutes after experimental food intake
Baseline subjective thirst | Baseline
  Visual analogue scale rating in a scale from 0 to 100 mm for the quantification of the perceived thirst before the experimental food intake at baseline
Postprandial subjective thirst | Up to 120 minutes
  Visual analogue scale ratings in a scale from 0 to 100 mm for the quantification the perceived thirst measured at 15, 30, 45, 60, 90 and 120 minutes after experimental food intake
Baseline blood glucose concentration | Baseline
  Blood glucose concentration before experimental food intake
Baseline blood insulin concentration | Baseline
  Blood insulin concentration before experimental food intake
Incremental area under the curve (iAUC) for glucose | 0,15,30,45,60,90,120
  The incremental area under the curve (AUCi) for glucose was calculated via the geometric sums of the areas of the triangles and trapezoids above the fasting glucose concentration over a 2-h period
Incremental area under the curve (iAUC) for insulin | 0,15,30,45,60,90,120
  The incremental area under the curve (AUCi) for insulin was calculated via the geometric sums of the areas of the triangles and trapezoids above the fasting insulin concentration over a 2-h period
Baseline blood high density lipoprotein cholesterol (HDL) concentration | Baseline
  Blood high density lipoprotein cholesterol (HDL) concentration before experimental food intake
Baseline blood low density lipoprotein cholesterol (LDL) concentration | Baseline
  Blood low density lipoprotein cholesterol (LDL) concentration before experimental food intake
Baseline blood triglyceride concentration | Baseline
  Blood triglyceride concentration before experimental food intake
Postprandial blood glucose concentration | Up to 120 minutes
  Blood glucose concentration measured at 15, 30, 45, 60, 90 and 120 minutes after the experimental food intake
Postprandial blood insulin concentration | Up to 120 minutes
  Blood insulin concentration measured at 15, 30, 45, 60, 90 and 120 minutes after the experimental food intake
Postprandial blood total cholesterol concentration | Up to 120 minutes
  Blood total cholesterol concentration measured at 15, 30, 45, 60, 90 and 120 minutes after the experimental food intake
Postprandial blood high density lipoprotein cholesterol (HDL) concentration | Up to 120 minutes
  Blood high density lipoprotein cholesterol (HDL) concentration measured at 15, 30, 45, 60, 90 and 120 minutes after the experimental food intake
Postprandial blood low density lipoprotein cholesterol (LDL) concentration | Up to 120 minutes
  Blood low density lipoprotein cholesterol (LDL) concentration measured at 15, 30, 45, 60, 90 and 120 minutes after the experimental food intake
Postprandial blood triglyceride concentration | Up to 120 minutes
  Blood triglyceride concentration measured at 15, 30, 45, 60, 90 and 120 minutes after the experimental food intake

CONTACTS AND LOCATIONS:
Overall Officials: Itziar Abete Goñi, PhD, Principal Investigator — Centre for Nutrition Research - University of Navarra; Santiago Navas Carretero, PhD, Principal Investigator — Centre for Nutrition Research - University of Navarra; M Ángeles Zulet Alzórriz, Professor, Study Director — Centre for Nutrition Research - University of Navarra; Carlos Javier González Navarro, PhD, Study Director — Centre for Nutrition Research - University of Navarra; J. Alfredo Martínez Hernández, Professor, Study Director — Centre for Nutrition Research - University of Navarra; Viviana Loria Kohen, PhD, Principal Investigator — IMDEA Food; Ana Ramirez Molina, PhD, Study Chair — IMDEA Food; Guillermo Reglero Rada, Professor, Study Chair — IMDEA Food; Elena Aguilar Aguilar, PhD, Study Chair — IMDEA Food; Helena Marcos Pasero, Study Chair — IMDEA Food; Susana Molina, Study Chair — IMDEA Food; Carmen Crespo, Study Chair — IMDEA Food; Cristina Galarregui Miquelarena, Study Chair — Centre for Nutrition Research - University of Navarra; Blanca Martínez de Morentín, MD, Study Chair — Centre for Nutrition Research - University of Navarra; Salomé Pérez Díez, Study Chair — Centre for Nutrition Research - University of Navarra; María Hernández Ruiz de Eguilaz, Study Chair — Centre for Nutrition Research - University of Navarra; Veronica Ciaurriz Fernández, Study Chair — Centre for Nutrition Research - University of Navarra; María Zabala Navó, Study Chair — Centre for Nutrition Research - University of Navarra; Begoña de Cuevillas García, Study Chair — Centre for Nutrition Research - University of Navarra; José Manuel Iniesta Chamorro, Study Chair — Universidad Politécnica de Madrid (UPM); Paloma Chausa Fernández, Study Chair — Universidad Politécnica de Madrid (UPM); José Tapia Galisteo, Study Chair — Universidad Politécnica de Madrid (UPM); Elena Hernando Pérez, Study Chair — Universidad Politécnica de Madrid (UPM); Enrique J. Gómez Aguilera, Study Chair — Universidad Politécnica de Madrid (UPM); Alexis Álvarez Rollán, Study Chair — Grupo I.C.A. Informática y Comunicaciones Avanzadas, S.L.; Alejandro García Rudolph, Study Chair — Institut Guttmann, University Institute attached to the Universitat Autònoma de Barcelona, Badalona, Barcelona, Spain; Universitat Autònoma de Barcelona, Bellaterra, Cerdanyola del Vallès, Spain; The Health Sciences Research Institute of the Germans; Alberto García Molina, Study Chair — Institut Guttmann, University Institute attached to the Universitat Autònoma de Barcelona, Badalona, Barcelona, Spain; Universitat Autònoma de Barcelona, Bellaterra, Cerdanyola del Vallès, Spain; The Health Sciences Research Institute of the Germans; Josep Maria Tormos Muñoz, Study Chair — Institut Guttmann, University Institute attached to the Universitat Autònoma de Barcelona, Badalona, Barcelona, Spain; Universitat Autònoma de Barcelona, Bellaterra, Cerdanyola del Vallès, Spain; The Health Sciences Research Institute of the Germans
Locations (1):
- Centre for Nutrition Research, University of Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Toro-Martin J, Arsenault BJ, Despres JP, Vohl MC. Precision Nutrition: A Review of Personalized Nutritional Approaches for the Prevention and Management of Metabolic Syndrome. Nutrients. 2017 Aug 22;9(8):913. doi: 10.3390/nu9080913. PMID 28829397
- [Background] Gonzalez-Muniesa P, Martinez JA. Precision Nutrition and Metabolic Syndrome Management. Nutrients. 2019 Oct 9;11(10):2411. doi: 10.3390/nu11102411. PMID 31601025
- [Background] Brooke, JB (1996). SUS - a quick and dirty usability scale. In: Usability Evaluation in Industry, Jordan, P, Thomas, B, Weerdmeester, B, and McLelland, I(eds), Taylor and Francis: London